CLINICAL TRIAL: NCT05180084
Title: Internet-administered Cognitive Behavioural Therapy for Young Adults With Low Self-esteem
Brief Title: Internet-administered CBT for Young Adults With Low Self-esteem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIYA
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-03

CONDITIONS: Self Esteem
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavior Therapy (Experimental): Therapist-Guided Internet based Cognitive Behavior Therapy
  Interventions: Behavioral: Cognitive behavior therapy
- Wait-list control (No Intervention): Wait-list control participants will receive the same treatment at the end of the study period.

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Internet-based CBT intervention based on CBT theory, self-determination theory and self-compassion therapy for low self-esteem among young adults.
  Arms: Cognitive Behavior Therapy

SUMMARY:
The study will investigate a CBT based treatment approach for low self-esteem among young adults.

DETAILED DESCRIPTION:
The study will test an adapted guided internet-delivered self-help program (Self-Esteem in Young Adults -SIYA) which lasts for seven weeks. Following recruitment via social media and a telephone interview, included participants will be randomized to active treatment or control. The control group will receive the intervention later.

ELIGIBILITY:
Inclusion Criteria:

Low self-esteem, as indicated by rating of < 20 the Rosenberg Self-Esteem Scale.

Age between 18 and 25 years old. Access to a computer, smartphone, or tablet with internet access. Write and speak Swedish. In case of use of psychotropical medication, a stable dose for the past three months prior to registration and no planned changes during the treatment.

Exclusion Criteria:

Other ongoing psychological treatment that affects the treatment received in the study.

No comorbid severe depressive symptoms and no suicidal plans. Ongoing alcohol use disorder, as indicated by Alcohol Use Disorders Identification Test (AUDIT).

Severe psychiatric comorbidities (e.g. psychosis, anorexia nervosa) that requires specialist care within the regular psychiatric care.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Change in Rosenberg Self-Esteem Scale | Before treatment, after 3 weeks, and after 7 weeks (post-treatment assesment).
  A 10-item measure of self-esteem. Sum scores range between 0-30. A higher score indicates a higher self-esteem.

SECONDARY OUTCOMES:
Change in Brunnsviken Brief Quality of Life Questionnaire | Before treatment and after 7 weeks (post-treatment assessment)
  Measure of subjective quality of life. Sum scores can range between 0 and 96. Higher scores indicate a higher quality of life.
Change in Robson Self-concept Questionnaire | Before treatment and after 7 weeks (post-treatment assessment)
  A 30-item measure of self-esteem. Sum scores range between 0-210. A higher score indicates a higher self-esteem.
Change in Self-Compassion Scale Short Format | Before treatment and after 7 weeks (post-treatment assessment)
  A 12-item measure of self-compassion. Sum scores range between 1-5. A higher score indicates higher self-compassion.
Change in Patient Health Questionnaire | Before treatment and after 7 weeks (post-treatment assessment)
  A 9 item measure of depressive symptoms. Sum scores range from 0-27. A higher score indicates more depressive symptoms.
Change in Generalised Anxiety Disorder 7-item scale | Before treatment and after 7 weeks (post-treatment assessment)
  Seven item measure of generalized anxiety disorder. Sum score range from 0 to 21, with higher scores indicating more generalized anxiety. Cut-offs for interpretation: 0-5 minimal anxiety, 6-9 mild anxiety, 10-14 moderate anxiety, and 15-21 severe anxiety.
Change in Alcohol Use Disorder Identification Test | Before treatment and after 7 weeks (post-treatment assessment)
  A 10 item measure of alcohol use disorders. Sum scores range from 0-40. A higher score indicates higher alcohol use.
Change in Performance based self-esteem Scale | Before treatment and after 7 weeks (post-treatment assessment)
  A 4-item measure of performance based self-esteem. Sum scores range between 4-20. A higher score indicates a higher performance based self-esteem.
Change in Rathus assertiveness schedule - 6 | Before treatment and after 7 weeks (post-treatment assessment)
  Six item measure of assertiveness. Sum score range from -18 to 18. A higher score indicates higher assertiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Principal Investigator — Linkoeping University
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No